CLINICAL TRIAL: NCT01072877
Title: A Randomized, Blinded, Multicenter Study to Evaluate the Efficacy and Safety of Polidocanol Injectable Foam 0.5%, 1.0%, or 2.0% Compared to Vehicle for the Treatment of Saphenofemoral Junction (SFJ) Incompetence
Brief Title: Efficacy and Safety Study of Polidocanol Injectable Foam for the Treatment of Saphenofemoral Junction (SFJ) Incompetence
Acronym: VANISH-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAP.VV015
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Varicose Veins
Keywords: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Polidocanol injectable foam 0.125% (Experimental): Polidocanol injectable foam 0.125%
  Interventions: Drug: Polidocanol injectable foam (PEM)
- Polidocanol injectable foam 0.5% (Experimental): Polidocanol injectable foam 0.5%
  Interventions: Drug: Polidocanol injectable foam (PEM)
- Polidocanol injectable foam 1.0% (Experimental): Polidocanol injectable foam 1.0%
  Interventions: Drug: Polidocanol injectable foam (PEM)
- Polidocanol injectable foam 2.0% (Experimental): Polidocanol injectable foam 2.0%
  Interventions: Drug: Polidocanol injectable foam (PEM)
- Vehicle (Placebo Comparator): Injection of vehicle comparator
  Interventions: Drug: Placebo Vehicle

INTERVENTIONS:
Drug: Polidocanol injectable foam (PEM) — Injection of Polidocanol injectable foam
  Arms: Polidocanol injectable foam 0.125%; Polidocanol injectable foam 0.5%; Polidocanol injectable foam 1.0%; Polidocanol injectable foam 2.0%
Drug: Placebo Vehicle — Placebo vehicle
  Arms: Vehicle

SUMMARY:
Varicose veins are enlarged, noticeably bulging veins, which commonly occur in the legs and may cause discomfort. In this study, patients with varicose veins in the legs will be participating. The purpose of this research study is to evaluate the safety and effectiveness of three different concentrations of an investigational drug, polidocanol injectable foam compared to vehicle (inactive solution) in treating the symptoms and appearance of varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* Incompetence of SFJ associated with incompetence of the GSV or other major accessory vein
* Ability to comprehend and sign an informed consent document and complete study questionnaires in English
* Ability to record symptoms in accordance with the protocol
* Symptomatic varicose veins
* Visible varicose veins

Exclusion Criteria:

* Patients who only have telangiectatic or reticular veins (Clinical Finding C1, as assessed by CEAP (clinical, etiologic, anatomic, and pathophysiologic) Classification of Venous Disorders).
* Leg obesity impairing the ability to access the vein to be treated and/or to apply postprocedure compression bandaging and stockings
* Ultrasonographic or other evidence of current or previous deep vein thrombosis or occlusion
* Deep vein reflux unless clinically insignificant in comparison to superficial reflux
* Peripheral arterial disease precluding the wearing of post-procedure compression bandaging and stockings
* Reduced mobility
* Major surgery, prolonged hospitalization or pregnancy within 3 months of screening
* Major co-existing disease (e.g. malignancy; pulmonary disease; renal or hepatic insufficiency; serious skin disease/condition that may compromise the ability of the patient to comply with the compression protocol, etc.)
* Known allergic response to polidocanol or heparin, including history of heparin-induced thrombocytopenia, and/or multiple allergic reactions
* Current alcohol or drug abuse
* Pregnant or lactating women
* Women of childbearing potential not using effective contraception
* History of DVT, pulmonary embolism or stroke

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Laguna Hills, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Bradenton, Florida
  - Oakbrook Terrace, Illinois
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Hartsdale, New York
  - New York, New York
  - North Tonawanda, New York
  - Stony Brook, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Toledo, Ohio
  - Bend, Oregon
  - Clarksville, Tennessee
  - Kirkland, Washington
  - Spokane, Washington

REFERENCES:
- [Derived] King JT, O'Byrne M, Vasquez M, Wright D; VANISH-1 Investigator Group. Treatment of Truncal Incompetence and Varicose Veins with a Single Administration of a New Polidocanol Endovenous Microfoam Preparation Improves Symptoms and Appearance. Eur J Vasc Endovasc Surg. 2015 Dec;50(6):784-93. doi: 10.1016/j.ejvs.2015.06.111. Epub 2015 Sep 16. PMID 26384639

RESULTS

PARTICIPANT FLOW:
Groups:
- Polidocanol Endovenous Microfoam 0.125%: Polidocanol endovenous microfoam 0.125%
  Polidocanol Endovenous Microfoam (PEM): Injection of Polidocanol Endovenous Microfoam
- Polidocanol Endovenous Microfoam 0.5%: Polidocanol endovenous microfoam 0.5%
  Polidocanol Endovenous Microfoam (PEM): Injection of Polidocanol Endovenous Microfoam
- Polidocanol Endovenous Microfoam 1.0%: Polidocanol endovenous microfoam 1.0%
  Polidocanol Endovenous Microfoam (PEM): Injection of Polidocanol Endovenous Microfoam
- Polidocanol Endovenous Microfoam 2.0%: Polidocanol endovenous microfoam 2.0%
  Polidocanol Endovenous Microfoam (PEM): Injection of Polidocanol Endovenous Microfoam
Period: Overall Study
Arm/Group | Vehicle | Polidocanol Endovenous Microfoam 0.125% | Polidocanol Endovenous Microfoam 0.5% | Polidocanol Endovenous Microfoam 1.0% | Polidocanol Endovenous Microfoam 2.0%
Started | 56 | 57 | 51 | 52 | 63
Completed | 55 | 56 | 51 | 50 | 63
Not Completed | 1 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Polidocanol Injectable Foam 2.0%: Polidocanol injectable foam2.0%
- Total: Total of all reporting groups
Arm/Group | Vehicle | Polidocanol Injectable Foam 0.125% | Polidocanol Injectable Foam 0.5% | Polidocanol Injectable Foam 1.0% | Polidocanol Injectable Foam 2.0% | Total
Number analyzed (Participants) | 56 | 57 | 51 | 52 | 63 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (11.31) | 51.6 (9.60) | 48.2 (11.78) | 48.8 (8.78) | 49.7 (10.49) | 48.9 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 42 | 37 | 38 | 47 | 208
  Male | 12 | 15 | 14 | 14 | 16 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 0 | 0 | 3
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 0 | 0 | 2
  Black or African American | 0 | 4 | 1 | 1 | 1 | 7
  White | 52 | 51 | 46 | 50 | 61 | 260
  More than one race | 0 | 2 | 2 | 1 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (5.95) | 28.8 (5.77) | 27.4 (5.75) | 28.6 (5.41) | 28.3 (5.40) | 28.2 (5.64)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-reported Symptoms of Varicose Veins (VVSymQ Score)
Description: The 9 varicose vein symptoms were to be assessed and graded on a 6-point (i.e., 0-5) duration scale and an 11-point (i.e., 0-10) intensity scale, and the patient's level of activity for that day was to be assessed and graded on the 6-point (i.e., 0-5) duration scale. The 9 varicose vein symptoms assessed using the e-diary were derived from the first question of the modified Venous Insufficiency Epidemiologic and Economic Study-Quality of Life/Symptoms (VEINES-QOL/Sym) instrument. The VVSymQ is a subset of 5 VEINESQOL/ Sym items that have been determined in earlier studies to be most important to patients (heaviness, achiness, swelling, throbbing, and itching).
  The daily VVSymQ score is the sum of the duration scores for these 5 symptoms (scores range from 0 to 25, with the lower end of the range being an indicator of less symptom intensity, and the higher end being an indicator of higher intensity).
  At Visit 2/baseline, Week 8, scores were calculated
Time Frame: Week 8
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Vehicle: Injection of vehicle
  Placebo Vehicle: Placebo vehicle
- Polidocanol Injectable Foam 0.125%: Polidocanol injectable foam at a 0.125% concentration
- Polidocanol Injectable Foam 0.5%: polidocanol injectable foam at a 0.5% concentration
- Polidocanol Injectable Foam 1.0%: Polidocanol injectable foam at 1.0% concentration
- Polidocanol Injectable Foam 2.0%: Polidocanol injectable foam at a 2.0% concentration
Arm/Group | Vehicle | Polidocanol Injectable Foam 0.125% | Polidocanol Injectable Foam 0.5% | Polidocanol Injectable Foam 1.0% | Polidocanol Injectable Foam 2.0%
Number analyzed (Participants) | 55 | 56 | 51 | 50 | 63
units on a scale | 2.13 (0.452) | 4.63 (0.447) | 5.68 (0.483) | 4.87 (0.477) | 5.78 (0.425)
Statistical Analysis 1: Comparison: Vehicle vs Polidocanol Injectable Foam 0.125%; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -2.49, 95% CI 2-sided [-3.72 to -1.27]
Statistical Analysis 2: Comparison: Vehicle vs Polidocanol Injectable Foam 0.5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.54, 95% CI 2-sided [-4.80 to -2.29]
Statistical Analysis 3: Comparison: Vehicle vs Polidocanol Injectable Foam 1.0%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-3.98 to -1.48]
Statistical Analysis 4: Comparison: Vehicle vs Polidocanol Injectable Foam 2.0%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.65, 95% CI 2-sided [-4.84 to -2.46]

2. Secondary Outcome: Change From Baseline to 8 Weeks in Appearance as Rated by Patient (PA-V3)
Description: The Patient Self-assessment of Visible Varicose Veins (PA-V3) instrument is a 5-point scale used by patients to evaluate the appearance of their visible varicose veins. On this single-item paper questionnaire, the instructions included a diagram of the medial view of a leg with the area between the ankle and the groin circled. The patient was instructed to choose 1 of 5 response options that best described the appearance of the visible varicose veins of the leg that was treated in the study. The patient was instructed not to consider the appearance of the leg outside the circled area or of any spider veins. Possible responses ranged from "Not at all noticeable" (a score of 0) to "Extremely noticeable" (a score of 4).
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Polidocanol Injectable Foam 1.0%: Polidocanol injectable foam at a 1.0% concentration
Arm/Group | Vehicle | Polidocanol Injectable Foam 0.125% | Polidocanol Injectable Foam 0.5% | Polidocanol Injectable Foam 1.0% | Polidocanol Injectable Foam 2.0%
Number analyzed (Participants) | 55 | 56 | 51 | 50 | 63
units on a scale | -0.15 (0.143) | -0.93 (0.142) | -1.40 (0.152) | -1.60 (0.151) | -1.75 (0.135)
Statistical Analysis 1: Comparison: Vehicle vs Polidocanol Injectable Foam 0.125%; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.17 to -0.40]
Statistical Analysis 2: Comparison: Vehicle vs Polidocanol Injectable Foam 0.5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-1.65 to -0.86]
Statistical Analysis 3: Comparison: Vehicle vs Polidocanol Injectable Foam 1.0%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-1.85 to -1.06]
Statistical Analysis 4: Comparison: Vehicle vs Polidocanol Injectable Foam 2.0%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.60, 95% CI 2-sided [-1.98 to -1.23]

3. Secondary Outcome: Change From Baseline at 8 Weeks Post Treatment in IPR-V3 Score- Physician Photographic Review of Appearance
Description: The Independent Photography Review - Visible Varicose Veins (IPR-V3) instrument is a 5-point scale used to assess the appearance of a patient's visible varicose veins. At baseline and Week 8, standardized digital photographs were taken of the medial view of the patient's target leg, from groin to ankle. An independent photography review panel, consisting of 3 trained, blinded clinicians evaluated the appearance of the patient's visible varicose veins using the IPR-V3 instrument's 5-point scale (where 0=none to 4=very severe visible varicose veins).
Time Frame: 8 weeks post treatment
Population: Population consists of all patients who had a baseline and on-treatment assessment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Polidocanol Injectable Foam 0.125% | Polidocanol Injectable Foam 0.5% | Polidocanol Injectable Foam 1.0% | Polidocanol Injectable Foam 2.0%
Number analyzed (Participants) | 55 | 56 | 51 | 49 | 61
units on a scale | -0.01 (0.081) | -0.46 (0.080) | -0.77 (0.086) | -0.76 (0.085) | -0.91 (0.077)
Statistical Analysis 1: Comparison: Vehicle vs Polidocanol Injectable Foam 0.125%; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.66 to -0.23]
Statistical Analysis 2: Comparison: Vehicle vs Polidocanol Injectable Foam 0.5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-0.98 to -0.53]
Statistical Analysis 3: Comparison: Vehicle vs Polidocanol Injectable Foam 1.0%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-0.97 to -0.53]
Statistical Analysis 4: Comparison: Vehicle vs Polidocanol Injectable Foam 2.0%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.11 to -0.68]

ADVERSE EVENTS:
Groups:
- Polidcanol Injectable Foam 0.5%: polidocanol injectable foam at a 0.5% concentration
- Polidocanol Endovenous Microfoam 2.0%: polidocanol injectable foam at a 2.0% concentration
Arm/Group | Vehicle | Polidocanol Injectable Foam 0.125% | Polidcanol Injectable Foam 0.5% | Polidocanol Injectable Foam 1.0% | Polidocanol Endovenous Microfoam 2.0%
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/57 | 0/51 | 0/52 | 0/63
Other Adverse Events (participants affected / at risk) | 20/56 | 38/57 | 46/51 | 41/52 | 50/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=56) | Polidocanol Injectable Foam 0.125% (N=57) | Polidcanol Injectable Foam 0.5% (N=51) | Polidocanol Injectable Foam 1.0% (N=52) | Polidocanol Endovenous Microfoam 2.0% (N=63)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 11 (11) | 10 (10) | 10 (10) | 6 (6)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 7 (7) | 5 (5) | 4 (4) | 8 (8)
Injection site hematoma (Vascular disorders) | 1 (1) | 3 (3) | 8 (8) | 4 (4) | 3 (3)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 6 (6)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 3 (3) | 6 (6) | 4 (4)
Injection site pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 3 (3)
Infusion site thrombosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 6 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 6 (6)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Edema peripheral (Vascular disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 3 (3)
Extravasation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No